CLINICAL TRIAL: NCT06870682
Title: Potential Effects of a Robot-based Upper Limb Rehabilitation Paradigm in Different Subgroups After Stroke: a Pilot Study
Brief Title: Potential Effects of Novel Sensorimotor Upper Limb Rehabilitation Paradigm
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Prof. Dr., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S69003; C2M/23/060 (Other Grant/Funding Number: KU Leuven)
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke; Upper limb; Sensorimotor; Sensory processing; Robot-based therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ROBUST intervention (Experimental): The participants will be measured a first time with both robot-based and clinical assessments. Thereafter, the participant follows a 4-week control period, only receiving standard care. After the control period, a second measuring moment is planned using the same outcome measures as during the first measurement. Then, a the 4-week intervention is planned, whereby participants get 48 hours additional sensorimotor upper limb training. They will come 3 times per week to Leuven for a therapy session of two hours. During these therapy sessions, they receive one hour robot-based therapy and one hour transfer package training with a therapist. Additionally, they follow 6 times a week a 1-hour home program. After this intervention period, they are measured a last time using the same outcome measures as during the previous measuring moments.
  Interventions: Behavioral: ROBUST

INTERVENTIONS:
Behavioral: ROBUST — During a 4-week intervention, participants get 48 hours additional sensorimotor upper limb training. They will come 3 times per week to Leuven for a therapy session of two hours. During these therapy sessions, they receive one hour robot-based therapy and one hour transfer package training with a therapist. Additionally, they follow 6 times a week a 1-hour home program. This intervention can be distinguished from others since it integrates both motor and sensory function, with focus on sensory processing. It combines robot-based therapy, a transfer package to daily activities, and a home program.

SUMMARY:
Sensorimotor function of the upper limb is often impaired after stroke, even in the chronic phase (minimum 6 months after stroke). Currently, an optimal intervention combining both motor and sensory function, with focus on sensory processing (one of the most important sensory functions), does not exists. However, the research team has developed a novel therapy paradigm combining robot-based training, a transfer package to daily life activities, and a home program. As a first step, the investigators will examine the feasibility and potential benefits of this novel therapy approach within this pilot study by recruiting 10 persons with chronic stroke. The investigators hypothesize that this therapy approach is feasible and potentially effective in chronic stroke.

DETAILED DESCRIPTION:
Sensorimotor function of the upper limb is often impaired after stroke, even in the chronic phase (minimum 6 months after stroke). Currently, an optimal therapy combining both motor and sensory function, with focus on sensory processing (one of the most important sensory functions), does not exists. However, the research team has developed a novel therapy paradigm combining robot-based training, a transfer package to daily life activities, and a home program. As a first step, the investigators will examine the feasibility and potential benefits of this novel therapy approach within this pilot study. This intervention study will recruit 10 persons with chronic stroke. The participants will be measured a first time with both robot-based and clinical assessments. Thereafter, the participant follows a 4-week control period, only receiving standard care. After the control period, a second measuring moment is planned using the same outcome measures as during the first measurement. Then, a the 4-week intervention is planned, whereby participants get 48 hours additional sensorimotor upper limb training. The participants will come 3 times per week to Leuven for a therapy session of two hours. During these therapy sessions, the participants receive one hour robot-based therapy and one hour transfer package training with a therapist. Additionally, the participants follow 6 times a week a 1-hour home program. After this intervention period, the particpants are measured a last time using the same outcome measures as during the previous measuring moments. The investigators hypothesize that this therapy approach is feasible and potentially effective in chronic stroke.

Optionally, if the participants is willing and able to, additional MRI and/or fNIRS assessments will be added to give a first idea regarding changes in brain structure, function and activity because of this novel therapy approach. This study will inform the investigators to finalize the protocol for a following RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures
2. A first-ever unilateral, supra-tentorial stroke, as defined by WHO (rapidly developing clinical signs of focal (or global) disturbance of cerebral function, with symptoms lasting 24 hours or longer or leading to death, with no apparent cause other than vascular origin)
3. ≥18 years old
4. Being in the chronic phase after stroke, i.e. > 6 months post stroke
5. Motor impairment in the upper limb, defined as Fugl-Meyer score >22 out of 66 to demonstrate moderate to full upper limb motor function (patients scoring <23 out of 66 will not be able to comply with the KINARM protocol)
6. Residual sensory upper limb impairment, defined as Tactile Discrimination Test score <24 out of 25
7. Impaired functionality, defined as Action Research Arm Test score <52 out of 57
8. Manageable spasticity for KINARM tasks

Exclusion Criteria:

1. Having musculoskeletal and/or other neurological disorders impacting care or prognosis
2. Having severe communication or cognitive deficits that interfere with the protocol
3. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the CIP
4. Contraindications for robot-based therapy (e.g., uncontrolled epilepsy)
5. Participation in another clinical investigation
6. Having uncontrolled head movements (e.g. tremor), only relevant if participant is willing to receive the additional fNIRS assessments
7. Having any contra-indications for MRI, only relevant if participant is willing to receive the additional MRI assessments:

   * Pacemaker
   * Implantable Cardioverter Defibrillator (ICD)
   * Cochlear implant
   * Internal Insulin-pump
   * Deep brain stimulation
   * Any other metal device in body
   * Claustrophobia
   * Having a history of a neuropsychiatric or neurologic disorder before the diagnosis of stroke (e.g., depression, traumatic brain injury)
   * Use of psychoactive medication before the diagnosis of stroke (e.g., anti-depressive medication)
   * Use (or history of use) of drugs/alcohol
   * Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-10-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test | From first measuring moment to last measuring moment after 8 weeks.
  Clinical assessment of motor activity performance on an ordinal scale ranging from 0 to 57, with higher scores meaning better performance

SECONDARY OUTCOMES:
Sensorimotor Action Research Arm Test | From first measuring moment to last measuring moment after 8 weeks.
  Clinical assessment of sensorimotor activity performance on an ordinal scale ranging from 0 to 57, with higher scores meaning better performance
Fugl-Meyer upper extremity assessment | From first measuring moment to last measuring moment after 8 weeks.
  Clinical assessment of motor function on an ordinal scale ranging from 0 to 66, with higher scores meaning better performance
Tactile discrimination test | From first measuring moment to last measuring moment after 8 weeks.
  Clinical assessment of sensory processing with an area under the curve based scoring system, with higher scores meaning better performance
Stroke Impact Scale | From first measuring moment to last measuring moment after 8 weeks.
  A self-report questionnaire that evaluates disability and health-related quality of life after stroke. A higher score indicates less disability and better quality of life.
Kinarm: Visually guided reaching task | From first measuring moment to last measuring moment after 8 weeks.
  Assessment of motor function using a 4-target centre-out reaching task on the Kinarm End-Point Lab
Kinarm: Arm position matching task | From first measuring moment to last measuring moment after 8 weeks.
  Assessment of limb position sense using a 9-target mirror-matching task on the Kinarm End-Point Lab
Kinarm: Passive and active discrimination task | From first measuring moment to last measuring moment after 8 weeks.
  Task on the Kinarm End-Point Lab used to assess passive and active sensory processing
Optionally: MRI assessment | From first measuring moment to last measuring moment after 8 weeks.
  MRI scan to study the structure and function of the brain.
Optionally: fNIRS assessment | From first measuring moment to last measuring moment after 8 weeks.
  The patient will be fitted with the fNIRS head cap during a standardized task on the Kinarm robot. This fNIRS measure studies brain activity during a sensorimotor activity.

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided